CLINICAL TRIAL: NCT07117370
Title: Assessing the Feasibility of Coach Mpilo for Men With TB and HIV in Eastern Cape, South Africa
Brief Title: Assessing the Feasibility of Coach Mpilo for Men With TB and HIV
Acronym: Coach Mpilo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34HL170819 (NIH); R34HL170819 (NIH)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coach Impilo (Experimental): Peer support for TB and HIV treatment
  Interventions: Behavioral: Coach Mpilo
- Standard of Care (No Intervention): Standard of care is treatment education and scheduled treatment pick up dates.

INTERVENTIONS:
Behavioral: Coach Mpilo — Peer support for treatment navigation. Peer supporters (coaches) with TB and HIV treatment experiences are trained in listening, support, and action planning to assist men in navigating and staying on treatment.
  Arms: Coach Impilo

SUMMARY:
Men are less likely to report TB-related symptoms, get diagnosed, smear convert, or complete treatment, suggesting that outcomes along the TB cascade are worse for men. Despite men's greater burden of TB and poorer treatment outcomes, no interventions have been developed to address these gendered disparities. Building on our preliminary research that identified men's preferences for a TB care support intervention, we identified Coach Mpilo (CM), a peer-support HIV treatment intervention that was developed by men for men in South Africa, and tailored for men TB infection. The aims of our study are to assess the feasibility of CM for men and assess secondary outcomes for treatment completion and HIV viral suppression to inform a Hybrid Type I intervention. In Aim 1, CM will be further tailored to men initiating TB treatment (CM-TB) and for with HIV co-infection (CM-TB/HIV). Using a mixed methods approach guided by ADAPT-IIT model, we will conduct interviews, CM simulations, and a pre-test to assess men's usability of CM-TB and CM-TB/HIV in this setting. We will conduct Aims 2 and 3 concurrently. In Aim 2, CM-TB will be evaluated to assess feasibility among men and secondary outcomes for retention in care and successful TB treatment (TBT) outcomes. Using a randomized controlled trial design, men (N=120) initiating TBT will be randomized to receive CM or clinic-based standard of care adherence support. The primary outcome is feasibility, acceptability, willingness and safety for men with secondary outcomes for completing TBT within 180 days per arm. In Aim 3, the feasibility of CM-TB/HIV for men (n=120) co-infected with TB and HIV will be assessed. The primary outcome is feasibility, acceptability, willingness and safety with secondary outcomes measured for proportion of men adherent to anti-retroviral therapy at TBT completion and with a suppressed viral (SVL) load 6 months post-ART initiation and post-TBT completion per study arm. If shown to be feasible, we will propose an randomized controlled trial to assess effectiveness in improving men's TB and HIV outcomes and adapted to improve men's health in the context of non-communicable diseases in South Africa and globally.

ELIGIBILITY:
Inclusion Criteria:

Aim 2: 1) men; 2) aged ≥18 years; 3) newly initiating (i.e., treatment naive) or re-initiating TBT after being loss-from-care per South African national guidelines; 4) live in BCM Health Districts; and 5) provide written informed consent.

Aim 3: 1) men; 2) aged ≥18 years; 3) newly initiating (i.e., treatment naive) or re-initiating TBT after being loss-from-care per South African national guidelines; 4) HIV-positive; 5) Not on ART, 6) live in BCM Health Districts; and 7) provide written informed consent.

Exclusion Criteria:

Aim 2: 1) Not a man; 2) aged < 18 years; 3) not initiating (i.e., treatment naive) or not re-initiating TBT after being loss-from-care per South African national guidelines; 4) not live in BCM Health Districts; and 5) cannot provide written informed consent.

Aim 3: 1) Not a man; 2) aged < 18 years; 3) not initiating (i.e., treatment naive) or not re-initiating TBT after being loss-from-care per South African national guidelines; 4) not HIV-positive; 5) on ART, 6) not live in BCM Health Districts; and 7) cannot provide written informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | From enrollment to the end of treatment and follow up at 180 days (Aim 2) From enrollment to the end of treatment and follow up at 210 days (Aim 3)
  Qualitative and quantitative assessment using interviews and surveys to evaluate intervention feasibility, acceptability, willingness and safety.

SECONDARY OUTCOMES:
TB treatment completion | From enrollment to intervention and follow-up at 180 days (Aim 2)
  Monthly medical record review of TB treatment pick-up.
HIV treatment | From enrollment to the end of intervention and follow-up at 210 days (Aim 3 only).
  Medical chart review of antiretroviral therapy pick-up and viral load.

CONTACTS AND LOCATIONS:
Locations (1):
- Desmond Tutu Health Foundation, East London, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daniels J, Medina-Marino A, Glockner K, Grew E, Ngcelwane N, Kipp A. Masculinity, resources, and retention in care: South African men's behaviors and experiences while engaged in TB care and treatment. Soc Sci Med. 2021 Feb;270:113639. doi: 10.1016/j.socscimed.2020.113639. Epub 2021 Jan 23. PMID 33493956
- [Result] Medina-Marino A, Bezuidenhout D, Ngcelwane N, Cornell M, Wainberg M, Beyrer C, Bekker LG, Daniels J. Qualitative Identification of Intervention Preferences to Support Men's Engagement and Retention in TB Care in South Africa. Am J Mens Health. 2022 Sep-Oct;16(5):15579883221129349. doi: 10.1177/15579883221129349. PMID 36218175
- [Result] Medina-Marino A, de Vos L, Daniels J. Social isolation, social exclusion, and access to mental and tangible resources: mapping the gendered impact of tuberculosis-related stigma among men and women living with tuberculosis in Eastern Cape Province, South Africa. BMC Glob Public Health. 2025 Jun 5;3(1):50. doi: 10.1186/s44263-025-00166-6. PMID 40474267